CLINICAL TRIAL: NCT03874364
Title: The Effect of Intraurethral Lidocaine Gel in Comparison With Plain Lubricating Gel on Pain Perception During Flexible Cystoscopy: A Prospective Randomized Study
Brief Title: The Effect of Intraurethral Lidocaine Gel on Pain Perception During Flexible Cystoscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ajet Hyseni (Other)
Responsible Party: Sponsor-Investigator, Ajet Hyseni, Dr.med.univ.RKS, Luzerner Kantonsspital
Organization: Luzerner Kantonsspital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Lidocaine-study
Record Dates: First submitted 2019-03-12; First posted 2019-03-14 (Actual); Last update posted 2019-03-14 (Actual); Status verified 2019-03

CONDITIONS: Flexible Cystoscopy
MeSH Terms: interventions — Counseling

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (8):
- Lidocaine gel, counselling, monitor (Active Comparator)
  Interventions: Device: Lidocaine gel; Other: Counselling; Other: Monitor
- Lidocaine gel, counselling, no monitor (Active Comparator)
  Interventions: Device: Lidocaine gel; Other: Counselling; Other: No monitor
- Lidocaine gel, no counselling, monitor (Active Comparator)
  Interventions: Device: Lidocaine gel; Other: Monitor; Other: No counselling
- Lidocaine gel, no counselling, no monitor (Active Comparator)
  Interventions: Device: Lidocaine gel; Other: No counselling; Other: No monitor
- Lubricating gel, counselling, monitor (Placebo Comparator)
  Interventions: Other: Counselling; Other: Monitor; Device: Lubricating gel
- Lubricating gel, counselling, no monitor (Placebo Comparator)
  Interventions: Other: Counselling; Device: Lubricating gel; Other: No monitor
- Lubricating gel, no counselling, monitor (Placebo Comparator)
  Interventions: Other: Monitor; Device: Lubricating gel; Other: No counselling
- Lubricating gel, no counselling, no monitor (Placebo Comparator)
  Interventions: Device: Lubricating gel; Other: No counselling; Other: No monitor

INTERVENTIONS:
Device: Lidocaine gel — 10 ml 2% lidocaine gel is instilled with a syringe through the length of the urethra and kept in site at least 5 minutes prior the introduction of the cystoscope.
  Arms: Lidocaine gel, counselling, monitor; Lidocaine gel, counselling, no monitor; Lidocaine gel, no counselling, monitor; Lidocaine gel, no counselling, no monitor
Other: Counselling — Patients receive a brochure in the waiting room explaining the procedure in details.
  Arms: Lidocaine gel, counselling, monitor; Lidocaine gel, counselling, no monitor; Lubricating gel, counselling, monitor; Lubricating gel, counselling, no monitor
Other: Monitor — Patients are allowed to view and follow the procedure on a monitor connected to the cystoscope's camera.
  Arms: Lidocaine gel, counselling, monitor; Lidocaine gel, no counselling, monitor; Lubricating gel, counselling, monitor; Lubricating gel, no counselling, monitor
Device: Lubricating gel — 10 ml plain lubrificant gel is instilled with a syringe through the length of the urethra and kept in site at least 5 minutes prior the introduction of the cystoscope.
  Arms: Lubricating gel, counselling, monitor; Lubricating gel, counselling, no monitor; Lubricating gel, no counselling, monitor; Lubricating gel, no counselling, no monitor
Other: No counselling — Patients won't receive a brochure in the waiting room explaining the procedure in details.
  Arms: Lidocaine gel, no counselling, monitor; Lidocaine gel, no counselling, no monitor; Lubricating gel, no counselling, monitor; Lubricating gel, no counselling, no monitor
Other: No monitor — Patients are not allowed to view and follow the procedure on a monitor connected to the cystoscope's camera.
  Arms: Lidocaine gel, counselling, no monitor; Lidocaine gel, no counselling, no monitor; Lubricating gel, counselling, no monitor; Lubricating gel, no counselling, no monitor

SUMMARY:
Flexible cystoscopy is routinely performed by urologists. Many patients have concerns to undergo this procedure and expect it to be unpleasant or even painful. Thus, reduction of pain and discomfort during cystoscopy is of great interest, but there is not sufficient evidence regarding the most appropriate conduct of cystoscopy.

In this study the impact of lidocaine gel, patient counseling and monitoring regarding pain perception during flexible cystoscopy are investigated.

ELIGIBILITY:
Inclusion Criteria:

* Men 18 - 80 years
* Given indication for flexible cystoscopy
* Written informed consent

Exclusion Criteria:

* Allergy to amid anesthetics
* Urinary tract infection
* Use of analgesics in the previous 24 hours and chronic intake of analgesics
* Dementia
* Presence of a sensory disorder such as or spinal cord injury
* Indwelling catheter carrier

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2021-01 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Pain based on a numeric rating scale | During flexible cystoscopy
  The pain scale ranging from 0 ("no pain") to 10 ("worst possible pain").

SECONDARY OUTCOMES:
Pain based on a numeric rating scale | Immediately before flexible cystoscopy
  The pain scale ranging from 0 ("no pain") to 10 ("worst possible pain").
Pain based on a numeric rating scale | 10 min after flexible cystoscopy
  The pain scale ranging from 0 ("no pain") to 10 ("worst possible pain").
Pain based on a numeric rating scale | 3 days after flexible cystoscopy
  The pain scale ranging from 0 ("no pain") to 10 ("worst possible pain").
Pain based on a verbal rating scale | Immediately after flexible cystoscopy
  The pain scale ranging from 0 ("it was not unpleasant") to 5 ("the investigation was almost unbearable").

CONTACTS AND LOCATIONS:
Locations (1):
- Klinik für Urologie, Kantonsspital Luzern, Lucerne, Switzerland